CLINICAL TRIAL: NCT02291172
Title: Comprehensive Communication Intervention for Minimally Verbal Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Ann Kaiser, Susan W. Gray Professor of Education and Human Development, Dept. of Special Education, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 141453
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention JEP (Experimental): A blend of JASP-EMT using SGDs with parent training intervention with the addition of individualized DTT to teach receptive language, imitation, and joint attention when children lack these skills at entry. The comprehensive communication intervention: (a) teaches foundational social communicative behaviors, (b) related skills that predict long term language outcomes, (c) a range of communicative functions, (d) spoken language skills, (e) provides children with an immediate mode of communication, (f) incorporates instructional methods, contexts, and partners that increase both the critical skills for spoken language and social use of language. Because parents are essential partners for young children with ASD who are learning to communicate, we (g) include parents
  Interventions: Behavioral: Intervention JEP
- Business as Usual Control Group (No Intervention): All children, regardless of group assignment will participate in all assessments. Children randomized to the control group will not receive intervention, but will complete all other research procedures. Other treatments that all children receive in the community will be recorded with bi-monthly surveys.

INTERVENTIONS:
Behavioral: Intervention JEP — A blend of JASP-EMT using SGDs with parent training intervention with the addition of individualized DTT to teach receptive language, imitation, and joint attention when children lack these skills at entry.
  Arms: Intervention JEP

SUMMARY:
Overview The goal of Comprehensive Communication Intervention for Minimally Verbal Children with Autism is to conduct an efficacy study of a promising intervention to increase spoken language in preschool children who are minimally verbal. The proposed study compares a comprehensive communication intervention (JASP- EMT Plus; JEP) to a business as usual (BAU) control group in a randomized controlled trial (RCT) across 4 time points. The study replicates and extends procedures used by Kasari, Kaiser et al (2014) to successfully promote social communication in older minimally verbal children. Intervention components include: (1) Joint Attention, Structured Play, Engagement and Regulation and Enhanced Milieu Teaching (JASP- EMT), (2) applied with systematic parent training, (3) use of speech generating device (SGD) and (4) supplementary direct teaching of foundational skills for language learning as indicated by child entry skills (CORE-DTT; Smith, 2009). Children who remain minimally verbal beyond age 5 are at high risk for persistent, severe communication deficits that impact social development, educational achievement and quality of life (Tager-Flusberg & Kasari, 2013). Thus, there is an urgent need for effective strategies to promote communication development during the preschool years to ameliorate early communication deficits and prevent persistent minimally verbal status. This study aims to change social communication in minimally verbal preschool children with ASD by applying a naturalistic social communication intervention which teaches the social foundations of communication and functional use of verbal language in play and interaction. In addition, the intervention addresses three factors that may contribute to remaining minimally verbal: lack of an effective mode of speech production, lack of foundational skills for learning language (receptive language, imitation, joint attention), and lack of communication partners to support continued language learning in natural environments.

DETAILED DESCRIPTION:
The proposed project is a randomized control design study testing the effectiveness of a comprehensive communication intervention to improve spoken language and social communication, and to reduce the portion of children with autism who are minimally verbal at age 5. The intervention (JASP-EMT-Plus; JEP) includes four components which have been shown to be effective in improving outcomes for older children with ASD who are minimally verbal. These components are (a) direct teaching for foundational language skills, (b) systematic introduction of an SGD paired with spoken language; (c) A naturalistic communication intervention: Joint Attention, Structured Play, Engagement and Regulation and Enhanced Milieu Teaching (JASP-EMT); and (d) parent training to support and generalize newly learned communication skills.

Following comprehensive assessment linking children's extant communication skills to the skills taught in each intervention component, an adapted treatment protocol will be developed for each child within the framework of the comprehensive treatment model. A total of 97 children ages 36 to 54 months will be randomly assigned to the treatment or a BAU control group. Progress in treatment will be monitored throughout the 3-month (42 session) intervention. Children will be assessed at 4 time points: pre intervention, post- intervention, 2 months, and 4 months after intervention. The data collected in this randomized trial will provide: (1) evidence of effectiveness for a comprehensive communicative intervention for improving communication in minimally verbal children with autism; and (2) new information about the correlates of minimal verbal status in children with autism.

Aim. To examine the effects of JEP on social communication (primary outcome) RQ1: Do young children with ASD who receive JEP produce significantly more social communicative utterances (proximal) in language samples, social communication on standardized assessment (distal), and expressive language on standardized assessment (distal) than children in the BAU group at T2 (immediately following intervention)?

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of ASD as confirmed by the ADOS
* Mental age (MA) of 18 months as measured on the Mullen Scales of Early Learning
* Expressive vocabulary of less than 10
* Age between 36 and 54 month
* English as the primary language spoken at home
* Parents who are willing to participate in parent training.

Exclusion Criteria:

* Exclusion criteria include any major medical conditions other than ASD, specifically a genetic disorders such as Down syndrome
* Sensory disabilities such as blindness or deafness
* Motor disabilities such as cerebral palsy.

Ages: 36 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Spontaneous communicative utterances | 12 weeks
  measured from a naturalistic language sample

CONTACTS AND LOCATIONS:
Locations (1):
- Metro Nashville Schools, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Hampton LH, Kaiser AP, Fuller EA. Multi-component communication intervention for children with autism: A randomized controlled trial. Autism. 2020 Nov;24(8):2104-2116. doi: 10.1177/1362361320934558. Epub 2020 Jul 6. PMID 32627570